CLINICAL TRIAL: NCT07342166
Title: Effect of Patellar Denervation on Post-operative Knee Pain and Knee Function in Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Effect of Patellar Denervation on Post-operative Knee Pain and Knee Function in Total Knee Arthroplasty
Acronym: PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 021/2566
Record Dates: First submitted 2025-12-25; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Patellar denervation; Total knee arthroplasty; Total knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patellar Denervation (Experimental)
  Interventions: Procedure: Patellar Denervation
- Non-Patellar Denervation (No Intervention)

INTERVENTIONS:
Procedure: Patellar Denervation — Electrocautery patella circumferentially during total knee arthroplasty
  Arms: Patellar Denervation

SUMMARY:
This study is a double-blind randomized controlled trial aiming to investigate the effects of patellar denervation using electrocautery on postoperative knee pain and knee function in patients undergoing primary total knee arthroplasty (TKA) without patellar resurfacing.

DETAILED DESCRIPTION:
This study is a prospective, double-blind randomized controlled trial conducted at Queen Savang Vadhana Memorial Hospital between 2023 and 2025. The aim of the study is to assess the effect of patellar denervation using electrocautery on postoperative knee pain and knee function in patients undergoing primary total knee arthroplasty (TKA) without patellar resurfacing.

Sixty-four patients were enrolled and randomly assigned to either the patellar denervation group (PD) or the non-denervation group (NPD), with 32 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-85 years old
* Knee osteoarthritis
* Plan for total knee arthroplasty after failed conservative treatment for at least 3 months

Exclusion Criteria:

* Previous history of trauma, fracture or open surgery on the same knee
* Inflammatory arthritis or Crystal-induced arthritis
* Patellar instability or isolated patellofemoral osteoarthritis
* Unable to answer questionnaire
* Cannot tolerate surgery due to medical comorbidities

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2025-06-21 (Actual)

PRIMARY OUTCOMES:
Visual analog scale score for knee pain | 2 weeks, 6 weeks, 3 months, 6 months, and 12 months

SECONDARY OUTCOMES:
Kujala score | 3 months, 1 year
Knee Society score | 3 months, 1 year
Timed up and go test | 3 months, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chalathorn Kulthonchalanan, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No
Data was save in form of Google sheet